CLINICAL TRIAL: NCT05996354
Title: A Study on the Concave Supra-arch Branched Stent-Graft System for Treatment of Aortic Arch Diseases
Brief Title: Concave Supra-arch Branched Stent-Graft System for Treatment of Aortic Arch Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJ-PR48-FIM-05
Record Dates: First submitted 2023-08-03; First posted 2023-08-18 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Aortic Dissection; Aneurysm, Aortic Arch; Aortic Pseudoaneurysm; Aortic Ulcer, Penetrating; Aortic Intramural Hematoma
MeSH Terms: conditions — Aortic Dissection; Aneurysm, Aortic Arch; Penetrating Atherosclerotic Ulcer; Aortic Intramural Hematoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Concave Supra-arch Branched stent-graft system
  Interventions: Device: Concave Supra-arch Branched stent-graft system

INTERVENTIONS:
Device: Concave Supra-arch Branched stent-graft system — To evaluate the efficacy and safety of the Concave Supra-arch Branched stent-graft system for endovascular treatment of aortic arch diseases.

SUMMARY:
There are no endoluminal stent systems available on the Chinese market for the effective treatment of aortic arch lesions (involving aortic arch aneurysms, aortic coarctation, aortic pseudoaneurysms, aortic ulcers, and intermural hematomas), and therefore this study is intended to be a prospective, single-arm study.

DETAILED DESCRIPTION:
The physician shall strictly follow the clinical study protocol and shall not deviate from or substantially change the protocol. However, in case of emergency such as immediate risk to the subjects, which needs to be eliminated immediately, it may be reported in written form afterwards. During the course of the study, documents such as amendments to the clinical study protocol and informed consent, requests for deviation, and resumption of the suspended clinical study shall be subject to the written approval of the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are ≥ 18 years old and ≤ 85 years old；
2. Patients with aortic arch diseases (involving aortic arch aneurysm, aortic dissection, aortic pseudoaneurysm, aortic ulcer, and intermural hematoma);
3. Anatomical criteria, including:

   1. Ascending aorta length is greater than or equal to 50 mm (distance from aortic sinus to anterior edge of innominate artery);
   2. The diameter range of the anchoring area at the proximal end of the main body is between 25-45 mm and the length is greater than or equal to 15 mm;
   3. The diameter of the anchored area of the innominate artery is between 10-16 mm, the diameter of the anchored area of the left common carotid artery is between 5-12 mm, and the diameter of the anchored area of the left subclavian artery is between 5-12 mm. Anchorage zone length is greater than or equal to 15 mm;
   4. Distance between the anterior edge of the innominate artery to the posterior edge of the left subclavian artery is less than or equal to 80 mm;
   5. Have a suitable iliac, femoral, and superior arch arterial approach;
4. Patients who understand the purpose of the study, volunteer to participate and sign the informed consent form, and are willing to complete follow-up visits as required by the protocol.

Exclusion Criteria:

1. Patients with general or local infections that may increase the risk of endovascular graft infection;
2. Patients with severe stenosis, calcification, or mural thrombus in the stent anchoring area, which is likely to make the stent-graft difficult to adhere to or affect the patency of the stent;
3. Patients with neck vascular surgery within 3 months;
4. Patients with severe carotid or subclavian artery stenosis, calcification;
5. Patients with a history of acute coronary syndrome within 6 months:

   Acute coronary syndromes are cardiac acute ischemic syndromes resulting from rupture of an unstable atherosclerotic plaque in the coronary artery or erosion secondary to the formation of new blood 4 thrombus, including ST-elevation myocardial infarction, non-ST elevation myocardial infarction, and unstable angina.
6. Patients with transient ischemic attack (TIA) or ischemic stroke within 3 months;
7. Patients with preoperative hepatic and renal dysfunction, [alanine aminotransferase (ALT) or aspartate aminotransferase (AST) exceeded the upper limit of normal level by a factor of five; Serum creatinine (Cr) >150umol/L];
8. Patients with history of bleeding or coagulopathy, who cannot receive antiplatelet therapy;
9. Patients with severe aortic insufficiency or a history of prior aortic valve insufficiency treatment;
10. Patients with a history of hypersensitivity to contrast agents, anticoagulant antiplatelet agents, stents, delivery equipment materials (i.e., nitinol, polyester, PTFE, nylon polymer materials);
11. Patients with connective tissue diseases such as Marfan's syndrome, Egyptian syndrome, or Behcet's disease;
12. Patients with arteritis;
13. Patients with significant organ dysfunction or other serious disease;
14. Patients with life expectancy of not more than 1 year;
15. Patients who are not eligible for endovascular treatment per in the investigator's judgment of the investigator;
16. Women with planned pregnancy, pregnancy stage , or lactation
17. The patient participated in another clinical trial and was not out or withdrawn within the first 3 months of the screening period of this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Immediate technical success rate | Immediate intraoperative
  Immediate technical success refers to the successful delivery system to a predetermined location, the successful deployment of the system and the safe withdrawal of the delivery system from the body, and the branch arteries were successfully reconstructed.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Chinese Academy of Medical Sciences Fuwai Hospital, Beijing, Beijing Municipality
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Yunnan Fuwai cardiovascular disease Hospital, YunNan, Yunnan

IPD SHARING:
Plan to Share IPD: No